CLINICAL TRIAL: NCT06857084
Title: Evaluation Of Clinical and Health Economic Outcomes Following Rotator Cuff Repair Using the REGENETEN◊ Bioinductive Implant: A Prospective, Multi-Center Global Registry
Brief Title: Evaluation Of Outcomes Following Rotator Cuff Repair Using the REGENETEN Bioinductive Implant: A Prospective, Multi-Center Global Registry
Acronym: RePaRe
Status: Recruiting | Type: Observational
Sponsor: Smith & Nephew, Inc. (Industry)
Collaborators: Smith & Nephew Asia Pacific Pte (Unknown)
Responsible Party: Sponsor
Other Study IDs: REGENETEN Global Registry
Record Dates: First submitted 2025-02-26; First posted 2025-03-04 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-01

CONDITIONS: Rotator Cuff Injuries
Keywords: Rotator Cuff Repair; Rotator Cuff Tear; Full Thickness Tear; Partial Thickness Tear; Massive Tear; REGENETEN Bioinductive Implant
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 7 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (1):
- Rotator cuff repair using REGENETEN: Patients undergoing arthroscopic rotator cuff repair using the REGENETEN Bioinductive Implant
  Interventions: Device: Arthroscopic rotator cuff repair with REGENETEN Bioinductive Implant augmentation

INTERVENTIONS:
Device: Arthroscopic rotator cuff repair with REGENETEN Bioinductive Implant augmentation — Arthroscopic rotator cuff repair aims at repairing the rotator cuff following tendon tear. The REGENETEN Bioinductive Implant is a medical device intended for the management and protection of tendon injuries. The REGENETEN Bioinductive Implant is indicated for the management and protection of rotator cuff tendon injuries in which there has been no substantial loss of tendon tissue.

SUMMARY:
This prospective, single-arm, multicenter registry is being conducted to collect real world post-market data from patients who are undergoing rotator cuff repair using the REGENETEN◊ Bioinductive Implant System. The Registry will include up to 50 centers in the United Kingdom (UK), Europe, Australia, and up to 400 patients for the initial evaluation.

Patients will be treated and evaluated according to standard medical care. Outcome data is collected up to 2 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject requires Arthroscopic rotator cuff repair (ARCR);
* Patients aged over 18 years old at the time of consent and providing baseline data before undergoing rotator cuff repair surgery (either partial or full thickness tears) will be eligible for this prospective registry.

Exclusion Criteria:

* Subject who, in the opinion of the Investigator, has an emotional or neurological condition that would pre-empt their ability or willingness to participate in the registry including mental illness, intellectual disability, and drug or alcohol abuse.
* Subjects who do not meet the indication or are contraindicated according to specific Smith+Nephew REGENETEN System's Instructions for Use (IFUs);
* Subject that meets the definition of a Vulnerable Subject per ISO14155:2020 Section 3.44.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Orthopaedic Clinics/practices
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2020-10-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
EuroQol 5 Dimension 5 Level (EQ-5D-5L) Score | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
  The descriptive system is used to describe the subject's health state & consists of 5 dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels to choose the most appropriate answer: no problems, slight problems, moderate problems, severe problems, and extreme problems. The subject is asked to indicate his/her health state by marking the most appropriate statement in each of the five areas. Responses are coded as single-digit numbers expressing the severity level selected in each dimension. For instance, 'slight problems' (e.g. 'I have slight problems in walking about') is always coded as '2'. The digits for the 5 dimensions are combined in a 5-digit code. The EQ- 5D-5L index value is derived by using the vendor supplied calculator to convert each 5-digit EQ-5D-5L profile. A higher number is a better outcome.
Quick DASH (Disabilities of Arm, Shoulder and Hand) Score | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
  Quick DASH (Disabilities of Arm, Shoulder and Hand) is designed to measure physical function and symptoms. It assesses 11 items, with scores ranging from 0 to 100 where 0 indicates no disability (i.e., better outcome) and 100 indicates most severe disability (i.e., worse outcome).
Oxford Shoulder Score (OSS) | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
  The Oxford Shoulder Score (OSS) is a questionnaire for the assessment of outcomes of shoulder surgery, which can reduce the observer's errors in the evaluation. It contains 12- item patient-reported outcome (PRO) measures specifically designed and developed for assessing outcomes of shoulder surgery such as assessing the impact on patients' quality of life of degenerative conditions (e.g., arthritis and rotator cuff problems).
  The OSS consists of 12 questions each scored 0 to 4 (0=unbearable, 1=severe, 2=moderate, 3=mild, 4=none) with 4 representing the best outcome. When the 12 items are summed, this produces overall scores that run from 0 to 48, with zero (0) representing a severe shoulder problem and 48 representing no related problem. Higher scores represent better clinical outcomes.
Pain, Visual Analog Scale (VAS) Score | Baseline, 2 weeks, 6 weeks, 3 months, 6 months, 12 months and 24 months
  Pain is assessed on a 100-point scale ranging from 0 to 100, with zero (0) representing no pain and 100 representing the worst pain imaginable
Single Assessment Numeric Evaluation (SANE) Score | Baseline, 6 weeks, 3 months, 6 months, 12 months and 24 months
  The Single Assessment Numeric Evaluation (SANE) is a simple but effective measure where patients rate their shoulder condition as a percentage (0-100%), where 100% being completely normal and 0% being the worst condition imaginable.

SECONDARY OUTCOMES:
Retear Rate | 3 months, 6 months, 12 months, and 24 months
  Cumulative 3 months, 6 months, 12 months, and 24 months retear rate. Failure is defined as Sugaya Type IV or V retear/recurrence (full-thickness discontinuity seen on both coronal and oblique sagittal MRI images).
Post-operative Recovery: Sling Type and Mobilization Time | 2 weeks
  The type of sling will be collected and presented for each treatment arm summarizing if standard sling, shoulder immobilizer, abduction sling, ER sling, or other were advised. Mobilization time will be calculated for both arms.
Post-operative Recovery: Return to Work | Baseline and 6 months
  Return to work questionnaires are collected at baseline and at 6 months post-op.
  At baseline, information on working arrangements are established:
  * Occupation status: Full time/part time/ retired
  * Occupation type: Sedentary/labor intensive
  * Impact of their diagnosis on their work performance: negative impact/no change
  At 6 months, information on changes to working arrangements is established:
  * Changes to occupation status
  * Returned to work and at what level: not returned due to procedure, not returned for other reasons, retired, lower level, same level, higher level
  * Time taken to return to work in days/weeks/months (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Scott Reid, Study Director — Smith & Nephew, Inc.
Locations (19):
- Melbourne Orthopaedic Group, Windsor, Victoria, Australia
- Clinique Saint Christophe, Soissons, Aisne, France
- Germany (6):
  - Schoen Klinik Lorsch, Lorsch, Rhine
  - Schoen Klinik Dusseldorf, Düsseldorf
  - Malteser Waldkrankenhaus Erlangen, Erlangen
  - Sporthopaedie Heidelberg, Heidelberg
  - St. Anna Hospital, Herne
  - OrthoMedicum Mittelhessen, Stadtallendorf
- Regional General Hospital F. Miulli, Acquaviva delle Fonti, Apulia, Italy
- United Kingdom (10):
  - Manchester University NHS Foundation Trust, Manchester, Greater Manchester
  - Spire Harpenden Hospital, Harpenden, Hertordshire
  - Spire Montefiore, Brighton, Hove
  - Burnley General Hospital, Burnley, Lancashire
  - Burnley General Teaching Hospital, Burnley, Lancashire
  - Manchester University NHS Foundation Trust, Manchester, Lancashire
  - Grantham and District Hospital, Grantham, Lincolnshire
  - University College London Hospitals, London, London
  - Cleveland Clinic London Hospital, London, London
  - Sulis Hospital Bath, Bath, Somerset

IPD SHARING:
Plan to Share IPD: No